CLINICAL TRIAL: NCT02677441
Title: Conservative or Surgical Management of Rockwood Type III to V Acromioclavicular Dislocations: A Non-inferiority Randomized Study
Brief Title: Conservative or Surgical Management of Rockwood Type III to V Acromioclavicular Dislocations
Acronym: AC Cons Chir
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: La Tour Hospital (Other)
Collaborators: Swiss Shoulder and Elbow Surgeons Expert Group (Unknown)
Responsible Party: Principal Investigator, Adrien Schwitzguebel, MD, La Tour Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GE 15-235
Record Dates: First submitted 2016-02-02; First posted 2016-02-09 (Estimated); Last update posted 2019-04-12 (Actual); Status verified 2019-04

CONDITIONS: Acromioclavicular Joint Dislocation; Conservative Versus Surgical Management
MeSH Terms: interventions — Conservative Treatment; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Conservative management (Experimental): Conservative management includes a sling for 10 days, followed by specific standardized validated rehabilitation that includes range of motion recovery and progressive reinforcement.
  Interventions: Procedure: Conservative management
- Surgery (Active Comparator): Surgical fixation of ACJD with coracoclavicular and acromioclavicular fixation, followed by specific standardized validated rehabilitation that includes range of motion recovery and progressive reinforcement.
  Interventions: Procedure: Surgery

INTERVENTIONS:
Procedure: Conservative management — Specific standardized rehabilitation protocol under Cote et al (2010)
  Arms: Conservative management
Procedure: Surgery — Coracoclavicular and acromioclavicular fixation as described ly Lädermann et al (2011), followed by specific standardized rehabilitation protocol under Cote et al (2010).
  Arms: Surgery

SUMMARY:
This study will evaluate the non-inferiority of conservative management for acromioclavicular clavicle disjunction, compared with surgical management. Half of patients will be treated with a specific standardized rehabilitation protocol, and the other half will be treated with coracoclavicular and acromioclavicular fixation, followed by a another specific standardized rehabilitation protocol.

Outcomes:

The primary outcome is the non-inferiority of the conservative management over surgical management of Rockwood III-V Acute acromioclavicular joint dislocation (ACJD) without PICCAT with American Shoulder and Elbow Surgeons (ASES score) at one year. If the non-inferiority is reached, the non-inferiority of the conservative management over surgical the management of Rockwood III-V ACJD with PICCAT using ASES score at one year will be evaluated.

Secondary outcomes were radiological criteria (i.e. comparison of ipsilateral and contralateral coracoclavicular distance on anterior view; and dynamic posterior shaft of the cross-body adduction Basamania/Alexander view) return to sports, work absenteeism, complication rate, cosmetic results, patients satisfaction, Constant score, Single Assesment Numeric Evaluation (SANE) score, Acromioclavicular Joint Instability (ACJI) score, ASES score at others timepoints, and range of motion of the implicated shoulder. Finally, multivariable regression analysis will be performed in order to evaluate the impact of predictors of interest on ASES score at one year.

DETAILED DESCRIPTION:
Background and rationale:

ACJD can be either managed conservatively or surgically. Concerning functional outcomes, it usually accepted that ACJD Rockwood state I and II should be treated conservatively.It is still debated whether grade III should be treated surgically or not, and only experts opinion suggest that grade IV and V has better surgical outcome than conservative. The main literature failed to demonstrate the superiority of the surgical management for functional outcomes. Despite this, operative management results in a better cosmetic outcome, but conservative management is associated with a lower duration of sick leave and lesser costs. It has been purposed by a worldwide expert consensus (ISAKOS consensus) that dynamic posterior clavicle impaction into the trapezius muscle (PICCAT) could be a predictive factor of poor functional outcome in case of conservative management.

Hypothesis:

H0: ASES score at one year of follow-up is better with surgical management than with conservative management.

H1: one year ASES score after conservative management is not inferior as after surgical management. H1 will be first tested without PICCAT. If H1 is validated, it will then be tested again including all patients, PICCAT or not.

Study design:

This multicentric case-control study is randomized 1:1 between conservative and surgical treatment of ACJD. It is a non-inferiority trial that includes 176 patients that suffers from acute ACJD Rockwood grade III-V. Conservative management will consist of a sling for 10 days followed by a standardized physical therapy program, (Cote et al. 2010) and surgical management will consist of coracoclavicular and acromioclavicular fixation and specific rehabilitation. Clinical follow-up will last one year.

Statistical analysis

Non-inferiority statistical analysis will be performed upon appropriate unilateral 95% confidence interval margin (Z = -1.645), with a non-inferiority margin of 6.4, corresponding to ASES minimal clinically important difference. Analysis is planned in case of "intention to treat" method, but, if patients of the conservative management group undergo surgery because they are unsatisfied, ASES score will be measured prior surgery instead of at one year of follow-up. No statistical adjustments on potential confounders are planned.

Sample size calculation:

ASES score minimal clinically important difference has been estimated to 6.4. ASES standard deviation after surgical management of ACJD has been estimated to 9.7. If there is truly no difference between the surgical and conservative treatments, then 80 patients are required to be 90% sure that the lower limit of a one-sided 95% confidence interval (or equivalently a 90% two-sided confidence interval) will be above the non-inferiority limit of -6.4. Mazzoca, one of the main authors of ISAKOS consensus (ISAKOS), has reported operating 50% of Rockwood type III-V ACJD. From this, we can strongly suppose that 50% of Rockwood type III-V ACJD presents PICCAT. Considering a 10% of drop-outs, we therefore need 80/(50%)*110% = 176 patients.

ELIGIBILITY:
Inclusion Criteria:

* acute (less than 10 days) ACJD , with possibility to perform surgery within 10 days after the trauma

Exclusion Criteria:

* Rockwood grade I, II, or IV ACJD
* Significant other trauma of the involved upper member requiring surgery
* Associated scapula or clavicle fracture
* Polytrauma inducing significant limitation of rehabilitation process
* Inability to follow properly conservative management or post-surgery recommendations
* Patients suffering from symptomatic anaemia, or patients with severe cardiorespiratory insufficiency
* Known or suspected non-compliance, drug or alcohol abuse
* Patients incapable of judgement or under tutelage
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc. of the participant
* Enrolment of the investigator, his/her family members, employees and other dependent persons

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Estimated)
Dates: Start 2016-02; Primary Completion 2021-12 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
The non-inferiority of the conservative management over surgical management of Rockwood III-V ACJD without PICCAT, regarding ASES score. | one year
The non-inferiority of the conservative management over surgical management of Rockwood III-V ACJD with and without PICCAT, regarding ASES score. | one year
  Will be considered as a secondary outcome if Outcome # 1 is not reached

SECONDARY OUTCOMES:
Coracoclavicular distance | one year
  Will be measured by comparing ipsilateral and controlateral X-ray
Dynamic posterior shaft of the clavicle | one year
  Will be measured on the cross-body adduction Basamania/Alexander view
Coracoclaviclular ligament integrity | one year
  Will be assessed on MRI, and scaled with grade 1 (tendinopathy), grade 2 (partial tear), and grade 3 (full tear) injury scale
Acromioclavicular ligament integrity | one year
  Will be assessed on MRI, and scaled with grade 1 (tendinopathy), grade 2 (partial tear), and grade 3 (full tear) injury scale
Return to sports | through study completion, an average of 1 year
Work absenteeism | through study completion, an average of 1 year
Complication rate | through study completion, an average of 1 year
cosmetic result | one year
  will be scaled on a visual analogue scale, from 0 to 10
patients satisfaction | one year
  will be scaled on a visual analogue scale, from 0 to 10
The non-inferiority of the conservative management over surgical management of Rockwood III-V ACJD without PICCAT, regarding Constant score. | 3, 6, and 12 months
The non-inferiority of the conservative management over surgical management of Rockwood III-V ACJD with and without PICCAT, regarding Constant score. | 3, 6, and 12 months
The non-inferiority of the conservative management over surgical management of Rockwood III-V ACJD without PICCAT, regarding ASES score. | 3, and 6 months
The non-inferiority of the conservative management over surgical management of Rockwood III-V ACJD with and without PICCAT, regarding ASES score. | 3, and 6 months
SANE score | 3, 6, and 12 months
ACJI score | 3, 6, and 12 months
pain VAS score | 3, 6, and 12 months
Range of motion: elevation of the involved shoulder | 3, 6, and 12 months
Ranges of motion: lateral rotation of the involved shoulder | 3, 6, and 12 months
Ranges of motion: medial rotation of the involved shoulder | 3, 6, and 12 months
Impact of predictors of interest on ASES score | one year
  Will be performed my multivariable regression analysis

CONTACTS AND LOCATIONS:
Overall Officials: Adrien Schwitzguébel, MD, Principal Investigator — La Tour Hospital
Locations (1):
- La Tour Hospital, Meyrin, Canton of Geneva, Switzerland

REFERENCES:
- [Background] Smith TO, Chester R, Pearse EO, Hing CB. Operative versus non-operative management following Rockwood grade III acromioclavicular separation: a meta-analysis of the current evidence base. J Orthop Traumatol. 2011 Mar;12(1):19-27. doi: 10.1007/s10195-011-0127-1. Epub 2011 Feb 23. PMID 21344264
- [Background] Tamaoki MJ, Belloti JC, Lenza M, Matsumoto MH, Gomes Dos Santos JB, Faloppa F. Surgical versus conservative interventions for treating acromioclavicular dislocation of the shoulder in adults. Cochrane Database Syst Rev. 2010 Aug 4;2010(8):CD007429. doi: 10.1002/14651858.CD007429.pub2. PMID 20687087
- [Background] Beitzel K, Mazzocca AD, Bak K, Itoi E, Kibler WB, Mirzayan R, Imhoff AB, Calvo E, Arce G, Shea K; Upper Extremity Committee of ISAKOS. ISAKOS upper extremity committee consensus statement on the need for diversification of the Rockwood classification for acromioclavicular joint injuries. Arthroscopy. 2014 Feb;30(2):271-8. doi: 10.1016/j.arthro.2013.11.005. PMID 24485119
- [Background] Cote MP, Wojcik KE, Gomlinski G, Mazzocca AD. Rehabilitation of acromioclavicular joint separations: operative and nonoperative considerations. Clin Sports Med. 2010 Apr;29(2):213-28, vii. doi: 10.1016/j.csm.2009.12.002. PMID 20226315
- [Background] Ladermann A, Grosclaude M, Lubbeke A, Christofilopoulos P, Stern R, Rod T, Hoffmeyer P. Acromioclavicular and coracoclavicular cerclage reconstruction for acute acromioclavicular joint dislocations. J Shoulder Elbow Surg. 2011 Apr;20(3):401-8. doi: 10.1016/j.jse.2010.08.007. PMID 20888260